CLINICAL TRIAL: NCT05271487
Title: The Effects of a Botanical Skin Care Regimen on Mild to Moderate Acne and the Microbiome
Brief Title: A Botanical Skin Care Regimen on Mild to Moderate Acne and the Microbiome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Integrative Skin Science and Research (Industry)
Collaborators: Codex Beauty Corporation (Unknown)
Responsible Party: Principal Investigator, Raja Sivamani, MD MS AP, Principal Investigator, Integrative Skin Science and Research
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CB_Acne_01
Record Dates: First submitted 2022-02-25; First posted 2022-03-09 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-02

CONDITIONS: Acne Vulgaris
Keywords: botanical; microbiome; skin care
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Multi-Step Botanical Skin Care Regimen (Experimental): The patient will be provided with and instructed to use a cleanser, toner, oil control cream, exfoliating facial scrub, clay mask, acne spot treatment, and body scrub for the duration of the study.
  Interventions: Other: Multi-Step Botanical Skin Care Regimen

INTERVENTIONS:
Other: Multi-Step Botanical Skin Care Regimen — The intervention includes 7 different topical products:
  1. Cleanser
  2. Toner
  3. Oil Control Cream
  4. Exfoliating Facial Scrub
  5. Clay Mask
  6. Acne Spot Treatment
  7. Body Scrub

SUMMARY:
The purpose of this study is to analyze changes in acne and changes in the gut and skin microbiome with the use of a multi-step botanical skin care regimen in those with mild to moderate acne.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 15 years of age until 45 years of age.
* The presence of mild to moderate acne based on investigator global assessment.

Exclusion Criteria:

* The presence of severe acne as noted by the investigator global assessment.
* Those with a nut allergy.
* Those who are unwilling to discontinue oral probiotic-based supplementation to meet the washout criteria prior to enrolling.
* Those who are unwilling to discontinue topical antibiotics and topical benzoyl peroxide to meet the washout criteria prior to enrolling.
* Individuals who are unwilling to discontinue vitamin E containing supplements during the washout and intervention.
* Individuals who have been on an oral antibiotic for acne within the previous 1 month.
* Individuals who are pregnant or breastfeeding.
* Individuals who have changed any of their hormonal based contraception within 3 months prior to joining the study.
* Oral supplementation that has nuts in it.
* Use of isotretinoin within the three months prior to joining the study.
* Current tobacco smoker or a tobacco smoking history of greater than 10 pack-years.

Ages: 15 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-03-07 (Estimated); Primary Completion 2022-07-01 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
Total lesion count | 8 weeks
  Number of of inflammatory lesions, and open and closed comedones

SECONDARY OUTCOMES:
Inflammatory lesion count | 4 weeks
  Number of inflammatory lesions
Inflammatory lesion count | 8 weeks
  Number of inflammatory lesions
Non-inflammatory lesion count | 4 weeks
  Number of open and closed comedones
Non-inflammatory lesion count | 8 weeks
  Number of open and closed comedones
Investigator global assessment (IGA) of acne | 4 weeks
  Validated scale for global assessment of acne. Scale is 0 to 4 with 4 indicating greater severity of acne
Investigator global assessment (IGA) of acne | 8 weeks
  Validated scale for global assessment of acne. Scale is 0 to 4 with 4 indicating greater severity of acne
Sebum excretion | 4 weeks
  Measure of skin sebum via sebumeter
Sebum excretion | 8 weeks
  Measure of skin sebum via sebumeter
Gut microbiome assessment | 4 weeks
  Gut microbiome shift for short-chain fatty acid producing bacteria via stool sample
Gut microbiome assessment | 8 weeks
  Gut microbiome shift for short-chain fatty acid producing bacteria via stool sample
Skin microbiome diversity | 4 weeks
  Shift in Shannon diversity of the skin microbiome
Skin microbiome diversity | 8 weeks
  Shift in Shannon diversity of the skin microbiome
Positive and Negative Affect Schedule (PANAS-SF) | 4 weeks
  Survey assessing positive and negative mood states. Scores range from 10 to 50 with higher scores representing positive affect
Positive and Negative Affect Schedule (PANAS-SF) | 8 weeks
  Survey assessing positive and negative mood states. Scores range from 10 to 50 with higher scores representing positive affect
Diurnal Cortisol Slope | 4 weeks
  4 salivary cortisol collections to assess diurnal slope
Diurnal Cortisol Slope | 8 weeks
  4 salivary cortisol collections to assess diurnal slope
Salivary Sex Hormone Levels | 4 weeks
  1 salivary collection to assess estradiol, progesterone, testosterone, DHEAS
Salivary Sex Hormone Levels | 8 weeks
  1 salivary collection to assess estradiol, progesterone, testosterone, DHEAS

CONTACTS AND LOCATIONS:
Locations (1):
- Integrative Skin Science and Research, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No